CLINICAL TRIAL: NCT04599751
Title: The Safety and Efficacy of Trio Diode Laser Module for Hair Removal Treatment in All Skin Types
Brief Title: The Trio Laser Module for Hair Removal Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alma Lasers (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALM-Trio-20-001
Record Dates: First submitted 2020-10-11; First posted 2020-10-23 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Hair Removal Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Hair removal treatment (Experimental): Trio laser module (Alma Lasers)
  Interventions: Device: Hair removal treatment

INTERVENTIONS:
Device: Hair removal treatment — Axilla and bikini line hair removal treatments using the Trio Laser Module (Alma Lasers).

SUMMARY:
The study is aimed to assess the safety and efficacy of hair removal treatments, using the Trio Laser Module (Alma Lasers).

The study will include 36 subjects that will undergo axilla and bikini line hair removal treatments. Safety and efficacy will be evaluated 3- months after the last treatment.

ELIGIBILITY:
Inclusion Criteria:

* Willing to undergo hair removal treatments at the Axilla and the Bikini line.
* Between 18 and 70 years of age.
* Reasonably good health, as defined by the Investigator.
* Agrees to avoid tanning during their participation in this study.
* Agrees to shave the treatment area prior to the treatment visit, according to the investigator's instructions.
* Subjects with dark brown hair.
* Eligible for treatment following a test spot without negative effects.
* Provided written Informed Consent and photo consent.

Exclusion Criteria:

* History of laser hair removal in the treatment area.
* Pregnant, lactating or planning to get pregnant within the study period.
* Unwilling to use a medically acceptable form of birth control at least 3 months prior to enrollment and during the entire course of the study, if of childbearing age.
* History of photosensitivity or use of medication with photosensitizing properties.
* Active infection in the treatment area.
* History or evidence of any chronic or reoccurring skin disease or disorder affecting the treatment area.
* History of keloid scarring or hypertrophic scar formation.
* Tattoo in the treatment area.
* Subject has been tanning within the past 30 days.
* History of confounding cancerous or pre-cancerous skin lesions in the treatment area.
* History of connective, metabolic or atrophic skin disease.
* Subject has used prohibited therapies, oral prescription medication, or topical meds (steroids) on the treatment area within 30 days prior to enrollment.
* History of autoimmune disorder

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2021-10-07 (Actual); Study Completion 2021-11-16 (Actual)

PRIMARY OUTCOMES:
Change in hair count | 3 month after the last treatment
  Change in hair count, preformed by blinded evaluators, based on photographs taken at 3m FU visit compared to baseline
Safety- Adverse events | Through study completion, an average of 1 year
  Adverse events and serious AE reported at any time during the trial or follow-up

SECONDARY OUTCOMES:
Investigator's assessment of the tolerability to the treatment using a 5-point Likert scale (when "0" indicates "none" and "4" indicates "sever"). | up to 24 weeks
  The investigator will assess the treatment area and score treatment related side effects using a 5-point likert scale, before and after the treatment
Subject's tolerability to the treatment, using a 5-point Likert scale (when "0" indicates "none" and "4" indicates "sever"). | up to 24 weeks
  Subjects will be requested to scale any sensation of stinging, tingling, itching and, burning using the 5-point Likert scale, before and after the treatment
Subject treatment related pain assessment, using VAS ( when "0" indicates "no pain" and "10" " worst possible pain" | up to 24 weeks
  Subjects will be requested to scale their treatment related pain
Subject's satisfaction from the treatment, using a 5-point Likert scale (when "1" indicates very dissatisfied and "5" very satisfied) | 3 months after the last treatment
  Subjects will be requested to scale their satisfaction from the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gold, MD, Principal Investigator — Tennessee Clinical Research Center; Edwardo Weiss, MD, Principal Investigator — Skin Care Research, LLC
Locations (2):
- United States (2):
  - Skin Care Research, LLC, Hollywood, Florida
  - Tennessee Clinical Research Center, Nashville, Tennessee